CLINICAL TRIAL: NCT06075407
Title: Evaluation of Fluid Resuscitation in Shocked Patients by Electrical Cardiometry in Comparison to Transthoracic Echocardiography
Status: Completed | Type: Observational
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abdel Aziz Abdel Raouf, Specialist of Anesthesiology, Surgical Intensive Care and Pain Medicine, Al-Azhar University
Other Study IDs: 0345/2023
Record Dates: First submitted 2023-10-04; First posted 2023-10-10 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Fluid Resuscitation; Electrical Cardiometry; Transthoracic Echocardiography; Shock
MeSH Terms: conditions — Shock

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fluid responder: All patients will undergo a volume expansion test or fluid challenge according to standard protocol. The volume expansion test will be performed with an intravenous infusion of 0.9% sodium chloride (500mL) within 15 minutes. The patient becomes a fluid responder if SV increases by > 10% after the fluid challenge.
  Interventions: Device: Assessment of fluid responsiveness by electrical cardiometry
- Fluid non-responder: All patients will undergo a volume expansion test or fluid challenge according to standard protocol. The volume expansion test will be performed with an intravenous infusion of 0.9% sodium chloride (500mL) within 15 minutes. The patient becomes a fluid responder if SV increases by > 10% after the fluid challenge (21). If the patient becomes a fluid non-responder, vasopressor infusion or inotrope will start.
  Interventions: Device: Assessment of fluid responsiveness by electrical cardiometry

INTERVENTIONS:
Device: Assessment of fluid responsiveness by electrical cardiometry — Electrical cardiometry (EC) measurements: by the ICON_ hemodynamic monitor (ICON Cardiotropic, Inc., La Jolla, CA 92307; Osyka Medical GmbH, Berlin, and Germany, model C3).
  Transthoracic echocardiography (TTE) measurements will be performed equipped with echo probe. SV of the left ventricle will be calculated using LVOT diameter (D) just below the aortic valve from parasternal long-axis view and VTI measured in LVOT from apical 5 chamber view (by pulsed wave Doppler).

SUMMARY:
The aim of this study is to evaluate the diagnostic accuracy of electrical cardiometry (EC) for the noninvasive determination of fluid responsiveness in critically ill shocked patients and agreement of EC compared to transthoracic echocardiography (TTE)

DETAILED DESCRIPTION:
Electrical cardiometry (EC), based on thoracic electrical bioimpedance, can measure SV continuously and non-invasively. The EC"s working principle of estimation of SV is to utilize changes in thoracic electrical impedance, which is mainly influenced by erythrocyte orientation and peak flow velocity in the ascending aorta throughout the cardiac cycle.

Electrical cardiometry (EC) has been validated to monitor SV and other hemodynamic parameters non-invasively compared to different techniques such as thermodilution technique, transesophageal Doppler echocardiography and cardiac catheterization including critically ill patients, intra-operative settings, in pregnant women, in children with congenital heart diseases, even in obese children

ELIGIBILITY:
Inclusion Criteria:

* Age from 25 to 65 years old.
* Both sexes.
* Patients with clinical criteria of shock [mean arterial pressure (MAP) ≤ 65 mmHg and tissue hypoperfusion (ScvO2 <70%, P(cv-a) CO2 ≥6 mmHg, CRT ≥4 s and lactate >2mmol/l).

Exclusion Criteria:

* Refusal to sign the consent by a first degree relative.
* Previous cardiac disease, rhythm other than sinus rhythm or heart rate > 140 beat/min.
* Renal failure (acute or chronic).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged from 25 to 55 years old were intubated, with clinical criteria of shock (mean arterial pressure (MAP) ≤ 65 mmHg).
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-04-29 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy of Electrical cardiometry (EC) to predict fluid responsiveness | Intraoperative and every 30 minutes till MAP>65mmHg
  Electrical cardiometry will be done be done immediately before fluid resuscitation and every 30 min till mean arterial pressure (MAP) > 65 mmHg

SECONDARY OUTCOMES:
Agreement of Electrical cardiometry(EC) with Transthoracic echocardiography (TTE) in the change of stroke volume before and after fluid challenge | Intraoperatively.
  Fluid resuscitation will be done by intravenous infusion of lactated ringer guided by fluid responsiveness (fluid responder if SV increases by > 10% after the fluid challenge. If the patient becomes fluid non-responder, vasopressor infusion or inotrope will start.
  The end of the study is when mean arterial pressure (MAP) > 65 mmHg (either by fluid or both fluid and vasopressor).

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.